CLINICAL TRIAL: NCT07048964
Title: A Prospective Cohort Study of Pralsetinib or Anlotinib in the Treatment of Locally Advanced and/or Metastatic Medullary Thyroid Carcinoma With RET Gene Mutations
Status: Not yet recruiting | Type: Observational
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: 22/284-3486
Record Dates: First submitted 2025-05-23; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Medullary Thyroid Cancer (MTC)
MeSH Terms: conditions — Carcinoma, Medullary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Drug: Pralsetinib
- Drug: Anlotinib

SUMMARY:
This trial is a prospective, observational Phase II clinical study. For patients with locally advanced and/or metastatic medullary thyroid carcinoma with RET gene mutations who require systemic treatment, they are randomly assigned to either the Pralsetinib or Anlotinib observation cohort based on their clinical treatment choices. The treatment continues until disease progression or the occurrence of intolerable adverse reactions. At the same time, the correlation between the efficacy and safety of the drugs and the RET gene mutation subtypes is analyzed, and the resistance mechanisms of Anlotinib and Pralsetinib are preliminarily explored to provide more evidence for the clinical treatment of patients with locally advanced or metastatic MTC in China.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Pathologically confirmed medullary thyroid carcinoma (MTC).
* Patients with locally advanced or metastatic MTC who require systemic treatment.
* Disease progression within 14 months before the screening visit.
* Presence of RET gene mutations based on tumor tissue and/or blood evaluations conducted by the study center.
* No prior treatment with pralsetinib and/or anlotinib and/or cabozantinib and/or vandetanib.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of 0-1.
* Expected survival time ≥ 3 months
* Signed informed consent to participate in this study.

Exclusion Criteria:

* The patient meets any of the following criteria within 14 days before the first administration of the study drug:

  1. Platelet count < 75 × 10^9/L.
  2. Absolute neutrophil count (ANC) < 1.0 × 10^9/L.
  3. Hemoglobin < 9.0 g/dL, with the possibility of elevating hemoglobin to 9.0 g/dL or higher through red blood cell transfusion and erythropoietin use, provided such treatment is completed at least 2 weeks before the first administration of the study drug.
  4. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 3 × upper limit of normal (ULN) without liver metastases; > 5 × ULN with liver metastases.
  5. Total bilirubin > 1.5 × ULN, > 3 × ULN with liver metastases; in the case of Gilbert's syndrome, total bilirubin > 3 × ULN and direct bilirubin > 1.5 × ULN.
  6. Estimated (Cockcroft-Gault formula) or measured creatinine clearance < 60 mL/min.
* The patient's QTcF > 470 msec. The patient has a history of long QT syndrome or torsades de pointes (TdP). The patient has a family history of long QT syndrome.
* The patient has clinically significant, uncontrolled cardiovascular diseases, including congestive heart failure classified as New York Heart Association (NYHA) Class III or IV; myocardial infarction or unstable angina within 6 months; uncontrolled hypertension; or clinically significant uncontrolled arrhythmias, including bradyarrhythmias that may lead to QT prolongation (e.g., second-degree atrioventricular block type II or third-degree atrioventricular block).
* The patient has metastatic central nervous system (CNS) tumors or primary CNS tumors with progressive neurological symptoms or requiring an increased dose of corticosteroids to control CNS disease. If corticosteroid treatment is needed for CNS disease, the dosing must be stable within the two weeks prior to C1D1.
* The patient has symptomatic interstitial lung disease or interstitial pneumonia, including radiation pneumonitis (i.e., affecting daily activities or requiring therapeutic intervention).
* The patient has received anti-tumor therapy within 14 days or five half-lives of the study drug prior to the first administration.
* The patient has received granulocyte colony-stimulating factor (G-CSF) support therapy within 14 days prior to the first administration of the study drug.
* The patient has undergone major surgery (excluding central venous catheterization, tumor biopsy, and gastrostomy tube insertion) within 14 days before the first administration of the study drug.
* The patient has been diagnosed with or requires treatment for another primary malignancy within the past 3 years, except for completely resected basal cell and squamous cell carcinoma of the skin, localized prostate cancer after curative treatment, and any in situ carcinoma that has been fully resected.
* The patient is unwilling or unable to comply with scheduled visits, dosing plan, laboratory tests, or other study procedures and restrictions.
* Non-menopausal or non-surgically sterilized female subjects are unwilling to use abstinence or highly effective contraception during the study drug administration and for at least 30 days after the last administration of the study drug; non-sterilized male subjects are unwilling to use abstinence or highly effective contraception during the study drug administration and for at least 90 days after the last administration of the study drug.
* Female patients who are currently breastfeeding.
* In the investigator's judgment, the patient has previous or current clinically significant conditions, medical history, surgical history, physical examination findings, or laboratory abnormalities that might affect patient safety, alter the absorption, distribution, metabolism, or excretion of the study drug, or interfere with the evaluation of study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with RET gene mutation-related locally advanced or metastatic medullary thyroid carcinoma (MTC) who require systemic treatment.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
To evaluate the objective response rate (ORR) of Pralsetinib or Anlotinib in patients with RET gene mutation-related locally advanced or metastatic medullary thyroid carcinoma (MTC) who require systemic treatment | 24 months
  Defined as complete response (CR) or partial response (PR) according to RECIST v1.1

SECONDARY OUTCOMES:
Progression-free survival (PFS) as assessed by Investigator | 24 months
Duration of Response (DOR) | 24 months
  Defined as the time from the first documentation of objective tumor response (CR or PR) to the first documentation of objective tumor progression or to death from any cause, whichever occurs first
Disease control rate (DCR) | 24 months
Changes in blood calcitonin (CT) and carcinoembryonic antigen (CEA) | 24 months
Safety: Type incidence and severity (as graded by NCI CTCAE v 4.0) of Pralsetinib or Anlotinib | 24 months
  Seriousness and attribution to the study medications of AEs and any laboratory abnormalities
Conversion rate of initially inoperable locally advanced medullary thyroid carcinoma (MTC) patients to surgically resectable status after treatment with pralsetinib or anlotinib | 24 months

OTHER OUTCOMES:
To explore the correlation of different RET gene mutation subtypes and other tumor tissue biomarkers with the efficacy and safety of drug treatment | 24 months
Preliminary exploration of resistance mechanisms in Chinese patients with locally advanced or metastatic RET-mutant medullary thyroid carcinoma (MTC) requiring systemic therapy after treatment with pralsetinib. | 24 months